CLINICAL TRIAL: NCT05542810
Title: A Prospective Randomized Trial to Compare the Effectiveness of Sports Drink and Water as a Solvent in Polyethylene Glycol for Colonoscopy
Brief Title: Compare the Effectiveness of Sports Drink and Water as a Solvent in Polyethylene Glycol for Colonoscopy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: GanHuoye (Other)
Responsible Party: Sponsor-Investigator, GanHuoye, Director of gastroenterology, Guangzhou Medical University
Organization: Guangzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Guangzhou Medical University
Record Dates: First submitted 2022-09-05; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Bowel Preparation

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sports drinks are polyethylene glycol solvents (Experimental)
  Interventions: Combination Product: Use sports drinks as polyethylene glycol solvents
- Water is a polyethylene glycol solvent (No Intervention)

INTERVENTIONS:
Combination Product: Use sports drinks as polyethylene glycol solvents — Using sports drinks as a polyethylene glycol solvent and water as a polyethylene glycol solvent in the control group, the effectiveness of intestinal preparation in the two groups was compared, and the adverse reactions, the acceptability of the solution taste, the timing of oral laxatives, and the willingness to repeat the same intestinal preparation or the willingness to recommend the same intestinal preparation to others were compared.
  Arms: Sports drinks are polyethylene glycol solvents

SUMMARY:
In this study, 200 patients were enrolled from 2023.1.1 to 2023.12.31, and were randomly divided into intervention and control groups. The intervention group compared the effectiveness of intestinal preparation in the two groups with sports drinks as a polyethylene glycol solvent and water as a polyethylene glycol solvent in the intervention group, and compared adverse reactions, acceptability of solution taste, time of oral laxatives, willingness to repeat the same intestinal preparation or the willingness to recommend the same intestinal preparation to others.

ELIGIBILITY:
Inclusion Criteria:

Hospitalized patients with gastrointestinal disorders Age 18 to 25 years

Exclusion Criteria:

Those who refuse to drink sports drinks Hypersensitivity to polyethylene glycol pregnant women, patients with suspected intestinal obstruction patients at risk of aspiration or with severe systemic or poorly controlled chronic disease patients with acute or severe disease and coagulation disorders patients with diabetes mellitus patients with a history of abdominal surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
A prospective randomized trial to compare the effectiveness of sports drink and water as a solvent in polyethylene glycol for colonoscopy | 1year
  After drinking, a questionnaire was used to compare the adverse reactions, acceptance, preparation time, and differences in the patient's willingness to prepare again or to recommend the same intestinal preparation method to others, and the results were expressed numerically.